CLINICAL TRIAL: NCT06138496
Title: Phase II Single-arm Clinical Study of the Efficacy and Safety of Cadonilimab in Combination With Lenvatinib Neoadjuvant Therapy for Patients With High-risk Renal Carcinoma Indicating Partial Nephrectomy
Brief Title: Cadonilimab Combination With Lenvatinib as Neoadjuvant Therapy for ccRCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, ZHOU FANGJIAN, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-117
Record Dates: First submitted 2023-11-13; First posted 2023-11-18 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cadonilimab; Clear Cell Renal Cell Carcinoma; Neoadjuvant Therapy
Keywords: Cadonilimab; Neoadjuvant therapy; Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cadonilimab combined with Lenvatinib as neoadjuvant therapy (Experimental): Lenvatinib Treatment Lenvatinib (8mg [body weight < 60 kg] or 12 mg [body weight ≥ 60 kg]) orally once daily, with or without food.
  Intravenous Infusion of Cadonilimab(Injection) Infuse Cadonilimab at a dose of 6mg/kg intravenously every two weeks, constituting one treatment cycle, a total of 3 or 6 cycles.
  Radical nephrectomy; Utilization of other targeted therapies; Combination targeted therapy with immunotherapy. If not, continue medication for three or six cycles before surgery.
  Interventions: Drug: Cadonilimab Combined With Lenvatinib

INTERVENTIONS:
Drug: Cadonilimab Combined With Lenvatinib — 3.7.1 Lenvatinib Treatment Lenvatinib (8mg [body weight < 60 kg] or 12 mg [body weight ≥ 60 kg]) orally once daily, with or without food.
  3.7.2 Intravenous Infusion of Cardonilli (Injection) Infuse Cardonilli at a dose of 6mg/kg intravenously every two weeks, constituting one treatment cycle, a total of 3 or 6 cycles.

SUMMARY:
Through the neoadjuvant treatment with a combination of Cardonilli and Lenvatinib, it enabled the successful and safe implementation of partial nephrectomy in patients with localized renal cancer, who had indications for nephron-sparing surgery but faced considerable difficulty in preserving the kidney (T1b with an endophytic component ≥75% or T2)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent (ICF).
2. Age ≥18 years old at the time of enrollment, male or female.
3. The Eastern United States Cancer Collaboration (ECOG) Physical Fitness score is 0 or 1.
4. Expected survival ≥3 months.
5. Preoperative biopsy pathologically confirmed clear cell carcinoma of kidney or renal cell carcinoma dominated by clear cell carcinoma
6. ECOG score 0 or 1
7. The patient has the intention of kidney preservation operation
8. There are indications for kidney-preserving surgery, but the operation is difficult (T1b endogenous ≥75% or T2).
9. Have at least one measurable lesion (according to mRECIST v1.1) suitable for repeated accurate measurement.
10. Good organ function, laboratory test results during the screening period meet the following criteria:

(1) Hematology (no use of blood components and cell growth factors to support therapy within 2 weeks before starting treatment) :

1. neutrophil absolute value (ANC) ≥ 1.5×109/L (1,500/mm3);
2. Platelet count (PLT) ≥ 100×109/L (100,000/mm3);
3. Hemoglobin (HB) ≥ 90 g/L; (2) Liver:

a. Serum total bilirubin (TBIL) ≤ 1.5×ULN; b. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) ≤ 2.5×ULN; For subjects with liver metastasis, AST and ALT ≤ 5×ULN c. Serum albumin (ALB) ≥28g/L (3) Coagulation function: International Standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN 11. Subject is willing and able to comply with scheduled visits, treatment protocols, laboratory tests, and other requirements of the study.

Exclusion Criteria:

* Lymph node metastasis
* Tumor surrounds renal artery
* Cancer thrombus in renal vein
* The tumor is diffuse and has no clear boundary with normal renal parenchyma
* Poor general status, anaesthetic assessment can not tolerate general anesthesia surgery
* Severe cardiovascular and cerebrovascular diseases, uncontrolled hypertension and diabetes
* Patients on long-term immunosuppressant use after organ transplantation
* Patients who are taking immunosuppressive drugs
* Patients with a definite infection or fever
* Patients with T-cell lymphoma and myeloma
* Patients who are combined with other malignant tumors, or are in the course of treatment for other benign and malignant tumors, or have a history of other malignant tumors within the past six months
* Metastatic kidney cancer.
* Received Chinese herbal medicines with anti-tumor indications or immunomodulatory effects within 14 days prior to the first use of the study drug
* Systematic therapy (including thymosin, interferon, interleukin, except for topical use to control pleural effusion).
* Have an autoimmune disease that is active or likely to recur, except for vitiligo, alopecia, psoriasis, or eczema that does not require systemic treatment; Hypothyroidism due to autoimmune thyroiditis requires only stable dose hormone replacement therapy; Only a steady dose of insulin replacement is required for type 1 diabetes.

Enrolling in another clinical study at the same time, unless it is an observational, non-interventional clinical study or follow-up period of an interventional study.

* Known history of mental illness, substance abuse, alcohol or drug use.
* Pregnant or breastfeeding women.
* The presence of any past or current medical condition, treatment, or laboratory test abnormality that may confuse the study results, interfere with the subject's full participation in the study, or that participation in the study may not be in the subject's best interest.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
ORR | Evaluation at the end of Cycle 3 or 6 (each cycle is 14 days) of Cadonilimab treatment
  Objective Response Rate (ORR) based on RECIST 1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No